CLINICAL TRIAL: NCT04160143
Title: Evaluating the Histologic Effects of Neoadjuvant Stereotactic Body Radiation Therapy (SBRT) Followed by Pulmonary Metastasectomy-Post SBRT Pulmonary Metastasectomy (PSPM) Trial
Brief Title: Post SBRT Pulmonary Metastasectomy (PSPM) Trial
Acronym: PSPM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SJHH_PSPM
Record Dates: First submitted 2019-10-29; First posted 2019-11-12 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-01

CONDITIONS: Surgical Resection; Stereotactic Body Radiotherapy; Lung Cancer; Pulmonary Metastasectomy
Keywords: Surgical resection; Stereotactic body radiation therapy; Pulmonary metastasectomy; Lung Cancers
MeSH Terms: conditions — Lung Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: This innovative study is an open-label unblinded single-arm prospective trial evaluating induction SBRT followed by pulmonary metastasectomy. As a Phase 2 trial, the primary purpose is to assess the efficacy of SBRT on metastatic tumor viability and the safety of SBRT as induction treatment prior to surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT followed by pulmonary metastasectomy (Experimental): SBRT+Surgery
  Interventions: Procedure: Surgical resection and stereotactic body radiation therapy (SBRT)

INTERVENTIONS:
Procedure: Surgical resection and stereotactic body radiation therapy (SBRT) — Surgical resection and stereotactic body radiation therapy (SBRT) are generally regarded as mutually exclusive treatment options for the local management of pulmonary malignancies. This Phase 2 prospective trial is a collaborative effort between the divisions of Thoracic Surgery and Radiation Oncology to evaluate the effects of dual treatment of pulmonary metastasis amenable to curative resection with neoadjuvant SBRT followed by surgical resection.

SUMMARY:
The goal of this study is to determine the effectiveness of SBRT on reducing tumor viability at a pathologic level and also to evaluate the effects of combined modality treatment on low volume pulmonary metastases, in hopes of extrapolating this information to both primary and secondary lung cancer.

DETAILED DESCRIPTION:
The role of SBRT as a potentially non-invasive treatment for small-volume tumors in the lung is well established, but the effectiveness of tumor eradication has yet to be determined. This prospective Phase 2 trial will provide several novel contributions to the literature: 1) the assessment of SBRT effectiveness in metastatic tumor control (radiotherapeutic metastasectomy), 2) the evaluation of pathologic response to SBRT by surgical resection, 3) identification of histologic predictors of radiation effect and toxicity (i.e. what are the effects of SBRT on different type of metastatic disease), and 4) the effect of combined modality SBRT and surgery on survival and local recurrence as compared to either modality alone. This trial will uniquely assess whether surgery as an adjunct to radiotherapy offers better tumor control as compared to SBRT alone, and whether it decreases locoregional recurrence. The study is an open-label unblinded single-arm prospective trial evaluating induction SBRT followed by pulmonary metastasectomy. This is a collaborative effort between the divisions of Thoracic Surgery and Radiation Oncology to evaluate the effects of dual treatment of pulmonary metastasis amenable to curative resection with neoadjuvant SBRT followed by surgical resection. Study recruitment and analysis will be conducted at St. Joseph Healthcare Hamilton and the Juravinski Cancer Center. Institutional data suggests that the Division of Thoracic Surgery at McMaster University performs an average of 450 pulmonary resections per year with approximately 10-15% being pulmonary metastasectomies for a spectrum of malignancies (including colorectal carcinoma, renal cell carcinoma and soft tissue sarcoma).

Surgical resection and stereotactic body radiation therapy (SBRT) are generally regarded as mutually exclusive treatment options for the local management of pulmonary malignancies. The Primary Outcome will be measured as the Rates of complete pathologic response (pCR) in surgical specimens post SBRT as assessed using the Junker grading scale for lung malignancies: Grade I, no regression or only spontaneous tumor regression; Grade II, morphologic evidence of tumor regression with at least 10% (grade IIa) or <10% (grade IIb) viable tumor tissue; and Grade III, complete tumor regression with no viable tumor. The Secondary Outcomes: Overall survival (OS) at 3 years, Disease-free survival (DFS) at 3 years, local recurrence rates, radiation related toxicity, postoperative pulmonary complication rate (including prolonged air leak, need for invasive or noninvasive mechanical ventilation, postop pneumonia and empyema), the effect on time-to-resection and tumour histology on pCR. In addition, it will be explored whether cancer specific tumor biomarkers correlate with SBRT effects and related toxicity. Based on institutional data from other local prospective trials, the Thoracic Surgery division at McMaster averages a study accrual rate of 25-30% and retention rate of approximately 80%. The most pertinent metric in determining the necessary sample size is the effect size estimate of pCR. The MISSILE study preliminary data demonstrated a pCR of 60%. This serves as the only representative value in the literature, even though our study evaluates SBRT and surgery for metastatic disease and NOT primary lung cancer. In contrast, the SBRT literature (using post-treatment CT scan surveillance only) reports local control rates of nearly 90%. Using the Fleming procedure, in order to measure the true pCR with a 95% confidence interval ± 10% using an estimated true pCR of 70%, estimated dropout rate of 20%, and 80% power, the calculated sample size requirement is 39 patients. It is estimated being able to recruit approximately 1-2 patients per month.

ELIGIBILITY:
Inclusion Criteria:

* Patient age >18, resectable pulmonary metastases without a more effective systemic therapy option (regardless of type of primary malignancy, excluding hematologic malignancies) with the primary malignancy already having been treated without evidence of local recurrence
* Patient having single-organ metastasis to lung only (with the exception of colorectal CA (Cancer) with synchronous hepatic metastasis)
* Tumors <5cm
* Patient with no evidence of nodal disease on pre-treatment CT scan
* Patient having adequate pulmonary function to tolerate lung resection (post-operative predictive FEV1≥40%).

Exclusion Criteria:• Patient having comorbidities not amenable to surgery

* Patient with uncontrolled primary malignancy
* Patient with hematologic malignancies (leukemia or lymphoma)
* Patient having more than 5 tumors in one lung
* Patient with prior history of thoracic radiation
* Patient having history of lung cancer diagnosis within 5 years of assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2020-07-14 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Rates of complete pathologic response (pCR) | post-operative 3 weeks
  pCR in surgical specimens post SBRT as assessed using the Junker grading scale for lung malignancies: Grade I, no regression or only spontaneous tumor regression; Grade II, morphologic evidence of tumor regression with at least 10% (grade IIa) or <10% (grade IIb) viable tumor tissue; and Grade III, complete tumor regression with no viable tumor.

SECONDARY OUTCOMES:
Overall survival (OS) | Post operative 3 years
  Followup over all survival (OS) at 3 years
Disease-free survival (DFS) | Disease-free survival (DFS) at 3 years
  Followup over all survival (OS) at 3 years. Based on 1. clinical 2. CT scan results
local recurrence rates | post operative 3 years
  CT scan at follow-up
Radiation related toxicity | Post radiation 1 year
  Follow Radiation Therapy Oncology Group (RTOG) Common Toxicity Criteria (Cox, 1995)
Postoperative pulmonary complication rate (including prolonged air leak, need for invasive or noninvasive mechanical ventilation, postop pneumonia and empyema) | post operative 30 days
  Using Society of Thoracic Surgery (STS) Database
The effect on time-to-resection and tumour histology on pCR | 8 to 12 weeks at different time post operative
  Time analysis
Identify mRNA tumor markers by Circulating Tumor Cell/CTC test | Baseline/ pre-SBRT; 6 Weeks post SBRT/6 weeks post Radiation , 6 weeks post Surgery
  Identify mRNA tumor markers for circulating tumor cell/CTC detection from blood sample to get cancer specific tumor biomarkers correlate with SBRT effects including different targeted gene such MUC1, HER2, EPCAM, ER/PR for Breast Cancer, PSA, PSMA, EGFR, AR for Prostate Cancer, EPCAM, EGFR, CEA for Colon Cancer, EPCAM, MUC1, CA125, ERCC1 for Ovarian Cancer and Stemcell . The CTC test will be doing to get information about whether or not disease has disseminated from the primary site and mainly as a prognostic and/or predictive marker in the metastatic settings. This test will be done in baseline or Pre SBRT, Post SBRT and Post Surgery.

CONTACTS AND LOCATIONS:
Overall Officials: John Agzarian, MD, MPH, Principal Investigator — McMaster University
Locations (1):
- McMaster University/St. Joseph's Hospital Healthcare, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang JY, Senan S, Paul MA, Mehran RJ, Louie AV, Balter P, Groen HJ, McRae SE, Widder J, Feng L, van den Borne BE, Munsell MF, Hurkmans C, Berry DA, van Werkhoven E, Kresl JJ, Dingemans AM, Dawood O, Haasbeek CJ, Carpenter LS, De Jaeger K, Komaki R, Slotman BJ, Smit EF, Roth JA. Stereotactic ablative radiotherapy versus lobectomy for operable stage I non-small-cell lung cancer: a pooled analysis of two randomised trials. Lancet Oncol. 2015 Jun;16(6):630-7. doi: 10.1016/S1470-2045(15)70168-3. Epub 2015 May 13. PMID 25981812
- [Background] Prezzano KM, Ma SJ, Hermann GM, Rivers CI, Gomez-Suescun JA, Singh AK. Stereotactic body radiation therapy for non-small cell lung cancer: A review. World J Clin Oncol. 2019 Jan 10;10(1):14-27. doi: 10.5306/wjco.v10.i1.14. PMID 30627522
- [Background] Ibrahim T, Tselikas L, Yazbeck C, Kattan J. Systemic Versus Local Therapies for Colorectal Cancer Pulmonary Metastasis: What to Choose and When? J Gastrointest Cancer. 2016 Sep;47(3):223-31. doi: 10.1007/s12029-016-9818-4. PMID 27080402
- [Background] Widder J, Klinkenberg TJ, Ubbels JF, Wiegman EM, Groen HJ, Langendijk JA. Pulmonary oligometastases: metastasectomy or stereotactic ablative radiotherapy? Radiother Oncol. 2013 Jun;107(3):409-13. doi: 10.1016/j.radonc.2013.05.024. Epub 2013 Jun 14. PMID 23773410
- [Background] Filippi AR, Guerrera F, Badellino S, Ceccarelli M, Castiglione A, Guarneri A, Spadi R, Racca P, Ciccone G, Ricardi U, Ruffini E. Exploratory Analysis on Overall Survival after Either Surgery or Stereotactic Radiotherapy for Lung Oligometastases from Colorectal Cancer. Clin Oncol (R Coll Radiol). 2016 Aug;28(8):505-12. doi: 10.1016/j.clon.2016.02.001. Epub 2016 Feb 18. PMID 26899780
- [Background] Junker K, Langner K, Klinke F, Bosse U, Thomas M. Grading of tumor regression in non-small cell lung cancer : morphology and prognosis. Chest. 2001 Nov;120(5):1584-91. doi: 10.1378/chest.120.5.1584. PMID 11713138
- [Background] Cox JD, Stetz J, Pajak TF. Toxicity criteria of the Radiation Therapy Oncology Group (RTOG) and the European Organization for Research and Treatment of Cancer (EORTC). Int J Radiat Oncol Biol Phys. 1995 Mar 30;31(5):1341-6. doi: 10.1016/0360-3016(95)00060-C. No abstract available. PMID 7713792
- [Derived] Begum H, Swaminath A, Lee Y, Fahim C, Bramson J, Naqvi A, Shargall Y, Finley C, Hanna W, Agzarian J. The histologic effects of neoadjuvant stereotactic body radiation therapy (SBRT) followed by pulmonary metastasectomy-rationale and protocol design for the Post SBRT Pulmonary Metastasectomy (PSPM) trial. Transl Cancer Res. 2022 Apr;11(4):918-927. doi: 10.21037/tcr-22-232. PMID 35571641